CLINICAL TRIAL: NCT04508101
Title: The Role of Suction Drainage in the Management of Peri-operative Bleeding in Total and Unicomcompartmental Knee Arthroplasty: a Comparative Retrospective Study
Brief Title: Suction Drainage in the Management of Peri-operative Bleeding in Total and Unicomcompartmental Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: DRGIN1
Record Dates: First submitted 2020-08-03; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Blood Loss, Surgical
Keywords: suction drainage; total knee arthtoplasty; unicompartmental knee arthroplasty
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- drainage group: Patients satisfying inclusion criteria who underwent either total as well as unicompartmental knee arthroplasty with suction drainage positioning
- non-drainage group: Patients satisfying inclusion criteria who underwent either total as well as unicompartmental knee arthroplasty without suction drainage positioning

SUMMARY:
Although, suction drainage is routinely used in orthopedic clinical practice, there are still no precise guidelines on its use in total joint arthroplasty, particularly in total as well as unicompartmental knee arthroplasty. In fact, drain use is likely associated to an increased risk of blood transfusion due to the lack of tamponade effect, as well as a higher infection rate. Furthermore, the drain itself could interfere with knee mobilization, delaying its functional recovery. Thus, the aim of this study was to investigate the real usefulness of suction drainage in perioperative bleeding control in the management of total as well as unicompartmental knee arthroplasty.

DETAILED DESCRIPTION:
Knee arthroplasty is currently a widespread treatment either for osteoarthritis (OA) as well as other joint disorders. Specifically, total knee arthroplasty (TKA) is commonly considered one of the most effective orthopedic procedure in the treatment of end-stage knee OA as well as various rheumatic diseases such as rheumatoid arthritis, leading to a substantial pain relief and functional improvement. Besides, unicompartmental knee arthroplasty (UKA) represents a viable alternative in the treatment of unicompartmental knee OA showing a lower morbidity. Nevertheless, since knee arthroplasty involves soft tissue dissections and numerous bone cuts, several perioperative complications can be observed. Particularly, the subsequent local hemorrhage can lead to anemia, functional limitation, nerve palsy as well as increase in wound tension resulting in healing impairment. Moreover, the local hematoma could represent a growth environment for bacteria. Although TKA usually shows a higher hemorrhage rate, some patients undergoing UKA still show the aforementioned complications. Accordingly, intraarticular suction drainage placement can likely ease the hematoma drain, leading to swelling decrease, surgical wound healing improvement as well as reduction of postoperative infections. However, despite suction drainage is routinely used in TKA as well as UKA, there are still no precise guidelines and its effectiveness remains controversial. Indeed, drain use is likely associated to an increased risk of blood transfusion due to the lack of tamponade effect, as well as a higher infection rate. Moreover, the drainage conduit could obstruct physiotherapy leading to a delayed recovery. Therefore, since fast-track program has been increasingly applied in the management of TKA and UKA, an early drainage removal is recommended. Thus, the aim of this study was to investigate the real usefulness of suction drainage in perioperative bleeding control in the management of TKA and UKA.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis diagnosis
* No contraindications to antithrombotic prophylaxis
* Availability of blood tests results before surgery as well as in the first three postoperative days.
* Detailed description of clinical records

Exclusion Criteria:

* contraindications to antithrombotic prophylaxis
* anti-platelet therapy
* knee arthroplasty revision indication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected from knee osteoarthritis with total as well as unicompartmental knee arthroplasty indication.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2020-08-07 (Estimated); Primary Completion 2020-08-24 (Estimated); Study Completion 2020-09-04 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin trend | 4 days
  Hemoglobin values comparison between the two groups

SECONDARY OUTCOMES:
Knee swelling | 5 days
  Evaluation of knee swelling during hospitalization (knee circumference variation > 2 cm)
Wound bleeding | 5 days
  Evaluation of wound bleeding during hospitalization (number of dressing changed)
Need for transfusion | 5 days
  Evaluation of transfusion rate during hospitalization (number of transfusions preformed)

CONTACTS AND LOCATIONS:
Overall Officials: Cristiana Balbino, MD, Principal Investigator — I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio

REFERENCES:
- [Derived] Manta N, Mangiavini L, Balbino C, Colombo A, Pandini EG, Pironti P, Vigano M, D'Anchise R. The role of suction drainage in the management of peri-operative bleeding in Total and Unicomcompartmental knee arthroplasty: a retrospective comparative study. BMC Musculoskelet Disord. 2021 Dec 10;22(1):1031. doi: 10.1186/s12891-021-04868-4. PMID 34893042